CLINICAL TRIAL: NCT04444648
Title: Longitudinal Evaluation of Circadian and Ultradian Rhythmic Fluctuations Measured by Continuous EEG During Coma to Predict the Recovery of Consciousness
Brief Title: Fluctuation of Rhymicity to Predict Recovery
Acronym: FR2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: FR2
Record Dates: First submitted 2020-05-25; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-05

CONDITIONS: Coma
MeSH Terms: conditions — Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One groupe without distinction of age, sexe, and pathology.: Patients with strok in coma, with or without wake up, and with disorder of consciousness. No limit in age (maybe give the younger age).
  We obtain this data from medical record. Every assessment was made of clinical purposes.
  We use the Glasgow coma recovery scale for assessment of behavior to check the variation of wakefulness. The scale was performed by the nursing staff every 2 to 8 hours depending on the severity of the medical condition.
  The continuous analysis of neurophysiologic data was based on EEG with a bipolar montage composed of the less noisy electrodes per recording period.
  The EEG features will include: spectral analysis (relative and absolute power in 4 canonical bands: Delta/Theta/Alpha/Beta) and complexity analysis (DFA, determinism, SVD entropy and permutation entropy).
  The patient outcome at the ICU and hospital discharges were collected from the medical files.
  Interventions: Combination Product: No intervention

INTERVENTIONS:
Combination Product: No intervention — No intervention

SUMMARY:
BRIEF SUMMARY :

In the most severe cases of brain injuries, intensive care may allow patients with altered consciousness to survive despite a significant risk of heavy sequelae. Persistent impairments of consciousness are currently categorized according to behavior in three main neurological categories: comatose state, vegetative state (recently named unresponsive wakefulness syndrome) and minimally conscious state. Refining the diagnosis of internal state is a major goal to determine the abilities for an optimal recovery of cognitive deficit. Circadian rhythms are implicated in the regulation of sleep-wake cycles but also in cognitive functions. Their role is actually revaluated in the mechanisms of consciousness impairment. First, it is well known that cognitive performances partially depend on such rhythms as they are more elevated during the day and correlated to the hormonal secretion. In a prognostic point of view, fewer rhythmic perturbations during the initial resuscitation period (with reorganized sleep rhythms and the presence of paradoxical sleep) could be associated to a higher functional outcome.

However, this internal state of alertness could be highly variable during the day as it might be influenced by specific rhythms such as the circadian rhythm. Only a continuous assessment could help defining them properly.

Thus, investigators hypothesize that the circadian restauration, assessed in a dynamic perspective, is associated with the improvement of content and level of awareness. The main challenge of our study is to capture the long-term changes in the evolution of circadian and ultradian rhythms and to keep a part of the natural history of the clinical recovery of these patients.

To achieve this goal, the investigators plan to analyze during more than 2 days both neurophysiological rhythms (EEG) and behavioral rhythms of alertness ("Eyes" scale from of the Glasgow coma scale) in a dataset collected retrospectively from the population of patients continuously monitored by EEG for medical purposes (to identify seizures and prevent status epilepticus) in an intensive care unit of teaching hospital as far as acquisitions last more than 48h and present no prolonged epileptic discharges or artifacts leading to uninterpretable EGG.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Admitted in ICU
* Altered level of consciousness not explained by a continuous sedation
* EEG during more than 48h consecutively

Exclusion Criteria:

* Prolonged epileptic discharges leading to uninterpretable EEG rhythms
* Prolonged artifacts leading to uninterpretable EEG trace

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose patient in ICU under intermittent behavioural evaluation and continuous EEG recording.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Status of awakening at the end of the period in the hospital | We analyze data obtained in a period between 2014 to 2017. The analysis is made since January 2020.
  The final outcome to assess the respective predictive value of behavioural assessment in ICU and EEG assessment of circadian and ultradian rhythms will be obtained by the medical record when the patient leave the hospital using a unique functional scale, namely the GOSE (Glasgow Outcome Scale - Extended).
  We use the Glasgow coma recovery scale for assessment of behavior to check the variation of wakefulness. The scale was performed by the nursing staff every 2 to 8 hours depending on the severity of the medical condition.
  The continuous analysis of neurophysiologic data was based on EEG with a bipolar montage composed of the less noisy electrodes per recording period.
  The patient outcome at the ICU and hospital discharges were collected from the medical files.

CONTACTS AND LOCATIONS:
Locations (1):
- Lyon teaching hospital, Hospices Civils de Lyon, Lyon, France